











## COVER PAGE WITH THE OFFICIAL TITLE OF THE STUDY:

Online Psychological Care Program To Reduce Psychological Distress In The Process Of Diagnostic Evaluation Of Mammary Glands In Women Who Attend A Breast Clinic.

**DATE: MARCH 21ST, 2023** 

## INFORMED CONSENT FOR THE ONLINE PSYCHOLOGICAL CARE PROGRAM TO REDUCE PSYCHOLOGICAL DISTRESS IN THE PROCESS OF DIAGNOSTIC EVALUATION OF MAMMARY GLANDS IN WOMEN WHO ATTEND A BREAST CLINIC.

Aimed at: Women undergoing diagnostic studies for breast cancer

Project title: Online psychological care program to reduce psychological discomfort in the process of diagnostic evaluation and/or screening of mammary glands in women who attend a breast clinic.

Name of the Principal Investigator: Dr. Reyna Jazmín Martínez Arriaga

You have been invited to participate in this research project, which is developed by members of the University Center for Health Sciences, the University of Guadalajara, the Technological Institute of Monterrey and the University of Twente, in coordination with the Mexican Social Security Institute.

If you decide to participate in the study, feel free to ask any questions that are not clear to you. It is important that you consider the following information:

The purpose of the present study is to evaluate the efficacy of an online psychological intervention to reduce anxiety, depression and negative psychological consequences and increase knowledge in patients undergoing their breast tests. The above, because it has been found in research that, in the diagnostic process of breast cancer, some women may present some psychological affectations. We ask you to participate in this study because you are part of the group of people who go to a breast clinic to get early detection tests for breast cancer.

You can enter the online psychological intervention through a virtual platform using an electronic device (cell phone, tablet, computer). In the platform you will find modules that contain short videos with psychological strategies that can help you in the process of carrying out your breast cancer detection studies.

To register on the platform, you will only be asked for an email and a password. Once you enter the platform, you will be asked to answer a series of questions to find out how you have been feeling in the last few days. These questions will be asked several times during the intervention, to assess the changes you are experiencing.

Your participation in this study may favor the area of research in health psychology, in order to improve health care in the Mexican population. On the other hand, it will not represent any cost to you.

Your identity and all the information that you provide us to enter the platform will be strictly confidential and will be used only by the research team of the project and will not be available for any other purpose. The results of this study may be published for scientific purposes, but will be presented in such a way that you cannot be identified.

Your participation in this study is completely voluntary. You are free to refuse to participate or to withdraw your participation at any time. Your decision to participate or not in the study will not imply any type of consequence in your care process at the breast clinic. If you agree to participate in the online psychological intervention, we ask you to click accept, otherwise you can close your Internet window. In this application, you inform that you agree to voluntarily participate in this research that we are conducting and, therefore, willing to complete the questionnaires.